CLINICAL TRIAL: NCT06956508
Title: Assessing the Impact of Prophylactic Targeted Brain Rehabilitation (TBR) on Phantom Limb Pain in the Perioperative Period Following Major Amputation, A Prospective Study
Brief Title: Prophylactic TBR on Phantom Limb Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: OrthoCarolina Research Institute, Inc. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HAND141
Record Dates: First submitted 2025-04-24; First posted 2025-05-04 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Phantom Limb Pain After Amputation
Keywords: Phantom Limb Pain; Targeted Brain Rehabilitation; VR; Virtual Reality
MeSH Terms: conditions — Phantom Limb

STUDY DESIGN:
Intervention Model Description: All Control Group patients will be retrospective subjects. Treatment Groups will be a single intervention enrolled prospectively.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): The control group will be any patients, 13 years old or older, who underwent major amputation with Dr. Gaston and Dr. Loeffler in 12-24 months before this trial started.
- Treatment Group (Active Comparator): The treatment group will be any patients, 13 years of age or older, who undergo major amputation with Dr. Gaston and Dr. Loeffler for 12-24 months after the start of the study.
  Interventions: Other: Targeted Brain Rehabilitation

INTERVENTIONS:
Other: Targeted Brain Rehabilitation — Patients will be given a virtual reality headset that is pre-loaded with the targeted brain rehabilitation (TBR) software at the time of their major amputation.
  The Virtual Reality (VR) environment will consist of a high-fidelity virtual representation of the participant's phantom limb. Participants will use a mounted head display (MHD) to interact with a virtual avatar, with the phantom limb represented as a realistic 3D limb model matching the remaining anatomy and skin tone. The VR system will be set up either in the clinic or at the participant's home, depending on individual circumstances and preferences.
  The VR protocol will be standardized and include exercises designed to mimic typical occupational therapy session.
  Arms: Treatment Group

SUMMARY:
This prospective study seeks to evaluate the effectiveness of prophylactic Targeted Brain Rehabilitation (TBR) in preventing or reducing Phantom Limb Pain (PLP).

DETAILED DESCRIPTION:
Phantom limb pain (PLP) affects 60-80% of amputees, including both upper and lower extremity amputees, leading to increased anxiety, depression, and reduced quality of life. With the total prevalence of major limb amputees in the United States projected to reach 3 million by 2050 and approximately 185,000 new cases annually, there is a pressing need for effective interventions to prevent and manage PLP.

Current pharmacologic treatments offer limited relief and can lead to adverse outcomes, particularly with long-term opioid use. Non-pharmacologic alternatives, such as mirror therapy, lack strong evidence supporting their efficacy and, to our knowledge, have not been evaluated in the perioperative period.

Virtual reality (VR) has emerged as a promising tool for mitigating various aspects of the phantom limb experience in major limb amputees. Previous research has shown that VR treatments can significantly reduce PLP, with many studies reporting a drop in numeric pain scores after VR use, and can be cost-effective. However, current literature on VR therapy for PLP has never evaluated its use in the immediate post operative period.

Initiating VR therapy immediately post-amputation may help in preventing maladaptive cortical reorganization, which is believed to be a key factor in the development of PLP. Following amputation, the sensory-motor cortex undergoes rapid rewiring as the brain attempts to compensate for the loss of sensory input from the amputated limb. This reorganization can lead to the formation of aberrant neural connections, contributing to the perception of phantom limb sensations and pain. By providing a virtual representation of the missing limb and facilitating its movement, VR therapy may be able to help maintain the integrity of the sensory-motor cortex, potentially preventing or reducing the development of PLP.

Our research team hypothesizes that prophylactic use of Targeted Brain Rehabilitation (TBR), a VR-based therapy system, in the perioperative period following major amputation can prevent or reduce the development of PLP and decrease the usage of opioids in this population. Furthermore, introducing VR therapy in the immediate post-operative period could help mitigate the psychological distress associated with amputation. By addressing both the physical and psychological aspects of amputation from the outset, prophylactic VR therapy has the potential to significantly improve the quality of life for amputees and reduce the long-term burden of PLP. Establishing the efficacy of prophylactic TBR in the perioperative period could revolutionize the standard of care for amputees, potentially reducing the incidence and severity of PLP and its associated psychological and quality of life impacts. This study will lay the groundwork for future multi-center, randomized controlled trials to validate the effectiveness of prophylactic TBR and establish it as a potential standard of care for amputees.

ELIGIBILITY:
Inclusion Criteria:

* 13+ year old patients undergoing major amputation with Dr. Gaston and Dr. Loeffler in the 12-24 months after the start of this study.
* Ability to read and comprehend English.
* Willing to use VR daily while in the inpatient setting following major amputation.

Exclusion Criteria:

* Patients under 12 years of age, and patients aged 13-17 without a legal guardian to give consent.
* Have used TBR extensively in the past for prior/unrelated amputation.
* Active uncontrolled mental illness
* Active neurological disease or cognitive impairment that would interfere with VR therapy or survey completion.
* Non-English speaking (surveys will only be provided in English)

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Short Form McGill Pain Questionnaire (SF-MPQ) | Through study completion, an average of 1 year
  Assesses quality/intensity of their pain experience using descriptive words. Consists of 15 descriptors rated on an intensity scale. Includes visual analog scale (VAS). Administered to both groups. One composite score.

SECONDARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | Through study completion, an average of 1 year
  Self-report pain on a scale of 0-10, where 0 means no pain and 10 means the worst pain imaginable
Brief Pain Inventory (BPI) - Short Form | Through study completion, an average of 1 year
  9-item questionnaire to assess pain severity and interference (two composite scores)
Phantom Limb Experience Survey | Through study completion, an average of 1 year
  Assesses presence, onset, location, character, intensity, triggers, and treatment of phantom limb sensations and phantom limb pain. Includes questions on phantom limb posture, movement, size changes, and telescoping.
Phantom Limb Assessment | Through study completion, an average of 1 year
  Assesses frequency, duration, and intensity of phantom limb pain compared to previous session. Assesses phantom limb posturing and control of phantom limb. Assesses duration of treatment effects in intervention group.
Simulator Sickness Questionnaire | Through study completion, an average of 1 year
  Assesses symptoms of simulator sickness including nausea, oculomotor problems, and disorientation. Only administered to intervention group.
System Usability Scale (SUS) | Through study completion, an average of 1 year
  Assesses subjective usability and satisfaction with the VR system. Scores range from 0 to 100, with higher scores indicating better usability.
Overall VR experience and feedback survey | Through study completion, an average of 1 year
  Supplemental questions to SUS
EuroQol five-dimensional health questionnaire (EQ-5D-5L) | Through study completion, an average of 1 year
  Assesses generic health status, quality of life, anxiety/depression
Patient Health Questionnaire-9 (PHQ-9) | Through study completion, an average of 1 year
  Objectifies and assesses degree of depression severity via questionnaire. Score ranges from 0 to 27, with higher scores indicating more severe depression.
Daily Pain Log - Additional Questions | Through study completion, an average of 1 year
  Assesses frequency and duration of phantom limb pain each day.

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Gaston, MD, Principal Investigator — OrthoCarolina Research Institute, Inc.
Locations (1):
- OrthoCarolina Research Institute, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rutledge T, Velez D, Depp C, McQuaid JR, Wong G, Jones RCW, Atkinson JH, Giap B, Quan A, Giap H. A Virtual Reality Intervention for the Treatment of Phantom Limb Pain: Development and Feasibility Results. Pain Med. 2019 Oct 1;20(10):2051-2059. doi: 10.1093/pm/pnz121. PMID 31165893
- [Background] Rothgangel, A. S., Braun, S., Schulz, R. J., Kraemer, M., de Witte, L., Beurskens, A., & Smeets, R. J. (2018). The PACT trial: patient centered telerehabilitation program for post-acute coronary artery disease patients. A prospective, multicenter, randomized controlled trial. Journal of Clinical Medicine, 7(10), 355.
- [Background] Rothgangel A, Braun S, Winkens B, Beurskens A, Smeets R. Traditional and augmented reality mirror therapy for patients with chronic phantom limb pain (PACT study): results of a three-group, multicentre single-blind randomized controlled trial. Clin Rehabil. 2018 Dec;32(12):1591-1608. doi: 10.1177/0269215518785948. Epub 2018 Jul 16. PMID 30012007
- [Background] MacIver K, Lloyd DM, Kelly S, Roberts N, Nurmikko T. Phantom limb pain, cortical reorganization and the therapeutic effect of mental imagery. Brain. 2008 Aug;131(Pt 8):2181-91. doi: 10.1093/brain/awn124. Epub 2008 Jun 20. PMID 18567624
- [Background] Wand BM, Parkitny L, O'Connell NE, Luomajoki H, McAuley JH, Thacker M, Moseley GL. Cortical changes in chronic low back pain: current state of the art and implications for clinical practice. Man Ther. 2011 Feb;16(1):15-20. doi: 10.1016/j.math.2010.06.008. Epub 2010 Jul 23. PMID 20655796
- [Background] Ambron E, Miller A, Kuchenbecker KJ, Buxbaum LJ, Coslett HB. Immersive Low-Cost Virtual Reality Treatment for Phantom Limb Pain: Evidence from Two Cases. Front Neurol. 2018 Feb 19;9:67. doi: 10.3389/fneur.2018.00067. eCollection 2018. PMID 29515513
- [Background] Vassantachart AY, Yeo E, Chau B. Virtual and Augmented Reality-based Treatments for Phantom Limb Pain: A Systematic Review. Innov Clin Neurosci. 2022 Oct-Dec;19(10-12):48-57. PMID 36591552
- [Background] Barbin J, Seetha V, Casillas JM, Paysant J, Perennou D. The effects of mirror therapy on pain and motor control of phantom limb in amputees: A systematic review. Ann Phys Rehabil Med. 2016 Sep;59(4):270-5. doi: 10.1016/j.rehab.2016.04.001. Epub 2016 May 30. PMID 27256539
- [Background] Alviar MJ, Hale T, Dungca M. Pharmacologic interventions for treating phantom limb pain. Cochrane Database Syst Rev. 2016 Oct 14;10(10):CD006380. doi: 10.1002/14651858.CD006380.pub3. PMID 27737513
- [Background] Von Korff MR. Long-term use of opioids for complex chronic pain. Best Pract Res Clin Rheumatol. 2013 Oct;27(5):663-72. doi: 10.1016/j.berh.2013.09.011. Epub 2013 Oct 5. PMID 24315147
- [Background] Ziegler-Graham K, MacKenzie EJ, Ephraim PL, Travison TG, Brookmeyer R. Estimating the prevalence of limb loss in the United States: 2005 to 2050. Arch Phys Med Rehabil. 2008 Mar;89(3):422-9. doi: 10.1016/j.apmr.2007.11.005. PMID 18295618
- [Background] Padovani MT, Martins MR, Venancio A, Forni JE. Anxiety, depression and quality of life in individuals with phantom limb pain. Acta Ortop Bras. 2015 Mar-Apr;23(2):107-10. doi: 10.1590/1413-78522015230200990. PMID 27069411
- [Background] van der Schans CP, Geertzen JH, Schoppen T, Dijkstra PU. Phantom pain and health-related quality of life in lower limb amputees. J Pain Symptom Manage. 2002 Oct;24(4):429-36. doi: 10.1016/s0885-3924(02)00511-0. PMID 12505212